CLINICAL TRIAL: NCT03293303
Title: The Feasibility, Effects and Costs of the 'Stay Active at Home Programme': Evaluation of a Preventive Integral Approach in Primary Care That Stimulates Physical Activity Among Community-dwelling Older Adults
Brief Title: The Feasibility, Effects and Costs of the 'Stay Active at Home Programme'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZonMw no. 50-53120-98-014
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Community-dwelling Older Adults
Keywords: Prevention; Physical activity; Sedentary behaviour; Daily activities; Homecare; Nursing; Primary care; Older adults; Function Focused Care; Reablement; Restorative Care
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with 12 months follow-up will be conducted. In total, five homecare teams from MeanderGroep Zuid-Limburg and the local domestic support workers will be trained in 'Stay Active at Home' (intervention group). Another five homecare teams and domestic support workers will deliver usual care (control group). Both groups of professionals and their clients will be compared at baseline and after 6 and/or 12 months follow-up.
Who Masked: Participant
Masking Description: Participants (i.e., older adults will be blinded); it's not possible to blind the healthcare professionals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stay Active at Home (Experimental): One group of homecare professionals receives a training programme. In this training they learn to motivate their clients to be more active in daily and physical activities.
  Interventions: Behavioral: Stay Active at Home
- Usual care (No Intervention): Second group of homecare professionals will get no training and their clients will receive usual homecare.

INTERVENTIONS:
Behavioral: Stay Active at Home — Stay Active at Home' aims to change the behaviour of community nurses and domestic support workers by offering them an intensive training programme. Subsequently, professionals are expected to deliver goal-oriented, holistic and person-centred services focusing on supporting older adults to maintain, gain or restore their competences to engage in physical and daily activities so that they can manage their everyday life as independently as possible.
  Arms: Stay Active at Home

SUMMARY:
BACKGROUND: Older adults spend approximately 80% of their awake time in sedentary activities which represents 8 to 12 hours per day. In the past, numerous stand-alone exercise programs have been developed. However, it is challenging to persuade older adults to become and maintain physically active. Consequently, physical activity should be embedded in the daily life of older adults to reduce their sedentary time, prevent negative health consequences and facilitate ageing in place.

INTERVENTION: 'Stay Active at Home' is not an additional, (classical) exercise programme; physical activity is integrated in usual home care. Healthcare professionals learn to engage older adults in daily life in order to improve their physical activity and reduce their sedentary time. For example, washing the upper body and face independently; changing the pillowcase, while professional changes bedcover; and motivating clients to join a dancing class at the community centre.

AIM and DESIGN: The aim of this cluster randomised controlled trial is to provide evidence about the (cost-) effectiveness of 'Stay Active at Home' prior to dissemination and implementation of the programme. Alongside the trial an extensive process evaluation will be conducted.

DETAILED DESCRIPTION:
Many community-dwelling older adults have a highly sedentary lifestyle, especially those receiving homecare services. In the Netherlands 20% of older adults makes use of homecare. The prevalence in frail older adults is even twice as high (40%). However, once in care often a downward spiral sets in, as professionals tend to meet their clients' needs by task completion rather than by stimulating self-management and active engagement in tasks to contribute to active ageing. Thereby they deprive older adults of their opportunities to engage in a routine range of movements necessary for maintaining underlying capability resulting in further deconditioning and functional decline.

To prevent these negative consequences the behaviour of healthcare professionals has to change from 'doing things for older adults' to 'engaging older adults' in daily life in order to improve physical activity among older adults by reducing their sedentary time. This innovative care philosophy is also known as Function Focused Care (FFC), restorative care or reablement. These terms can be used interchangeably, but we will refer to it as FFC throughout this project proposal. In the US the research group of Resnick and colleagues conducted various studies in inpatient and residential care facilities. They have shown that FFC succeeds in increasing physical activity. Furthermore, FFC has shown to result in physical (e.g. daily functioning, muscle strength, balance) and psychological benefits (e.g. mood, behavioural symptoms) and reduces the risk for adverse outcomes (e.g. falls, delirium). Resnick et al. have little experience in homecare settings, but there is an emerging body of evidence, especially in Norway, New Zealand and Australia, that FFC has also potential for community-based care showing beneficial effects with regard to daily functioning, self-perceived activity performance and satisfaction, health-related quality of life, healthcare utilisation/costs, and even mortality. Experiences and results of FFC in Dutch community-dwelling older adults are lacking.

Promising programmes in one particular care setting are not automatically replicable in other settings due to cultural or organisational differences. Consequently, available programmes need to be adapted to the local circumstances before they can be successfully implemented in another setting. However, making changes requires careful planning and execution to prevent a loss of effectiveness by affecting the original programme's theory or removing core components of the programme. Therefore, the investigators have followed so far the first two phases of the framework of the Medical Research Council in preparing the use of FFC in Dutch community-dwelling older adults receiving homecare services:

* Phase I (2013- first half of 2016): The investigators systematically adapted in co-creation with international FFC experts and a Dutch panel of relevant stakeholders the initial FFC philosophy and conducted a pilot study. Throughout the adaptation process healthcare professionals, policy makers, managers and scientists were involved at various times to ensure that all interests are considered and respected. Although not the primary target population (i.e. homecare professionals), the project idea was also intensively discussed with a panel of older adults. The final result of this adaptation process was the 'Stay Active at Home' programme (in Dutch: 'Blijf Actief Thuis'). During the pilot, data about its feasibility was collected from healthcare professionals and older adults.
* Phase II (second half of 2016 - first half of 2017): The investigators conducted a second pilot study, a so-called 'early trial' prior to the currently proposed trial, as part of the ZonMw project BASIC CARE REVISITED (ZonMw #520002003). This early trial provided relevant information regarding: a) the implementation of specific intervention components; b) key components of the chosen methodology (e.g. outcome measures); c) rates of recruitment and retention; and d) the expected effect size. This information is highly relevant with regard to finalising the intervention and designing a subsequent main trial.

In conclusion, 'Stay Active at Home' is systematically developed for the Dutch homecare setting based on international evidence in close collaboration with Dutch stakeholders (i.e. older adults, healthcare professionals, policy makers and managers). The initial feasibility of the programme and the proposed study design are evaluated in two pilot studies prior to the grant period. In order to determine the (cost-) effectiveness of 'Stay Active at Home' prior to dissemination and implementation of the programme in the Dutch homecare setting this cluster randomised controlled trial has to be conducted. Alongside the trial an extensive process evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Receive home care services by the selected nursing teams
* Age ≥65 years

Exclusion Criteria:

* Terminal ill or bedbound
* Serious cognitive or psychological problems
* Not able to communicate in Dutch

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 265 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Sedentary behaviour measured by ActiGraph GT3X+ (older adults) | 12 months
  An accelerometer that measures sedentary time and physical activity by assessing the magnitude of the body's acceleration in terms of 'counts' per unit time.

SECONDARY OUTCOMES:
Disabilities in ADL and IADL by Groningen Activity Restriction Scale (older adults) | baseline and after 12 months
  The Groningen Activity Restriction Scale (GARS) is a non-disease-specific instrument to measure disability in activities of daily living (ADL) and instrumental activities of daily living (IADL). For each item, four hierarchical answer options are available ranging from 'Yes, I can do it fully independently without any difficulty' to 'No, I cannot do it fully independently. I can only do it with someone's help'. The scores for the total scale range from 18 to 72, with higher scores indicating more disability
Physical activity by Short Physical Performance Battery (older adults) | baseline and after 12 months
  The Short Physical Performance Battery (SPPB) is a performance-based test of lower extremity function designed for elderly participants. It consists of three parts: the Balance Test, the Gait Speed Test, and the Chair Stand Test.Each test is scored 0 to 4 by previously determined criteria. Scores from the three tests will be summed into a composite score ranging from 0 to 12, with higher scores reflecting better physical functioning.
Major and minor depression by Patient Health Questionnaire-9 (older adults) | baseline and after 12 months
  The PHQ-9 is the first self-report questionnaire designed for use in primary care that reflects the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnostic criteria for depression, and so (through examining the pattern and number of items endorsed) can be used as a diagnostic tool for major and minor depression. The PHQ-9 consists of nine items which measure the presence of depressive symptoms. Participants will score how often each of the symptoms was present during the last two weeks (0 = not at all; 1 = several days; 2 = more than half of the days; 3 = nearly every day). The summary score ranges from 0 to 27, with higher scores reflecting more severe symptoms of depression.
Falls, 1 item 'How often did you fall during the last 6 months?' (older adults) | baseline and after 6, 12 months
  One item about falls
Health-related quality of life by EQ-5D-5L (older adults) | baseline and after 6, 12 months
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The EQ-5D-5L has 5 levels of severity for each of the 5 dimensions, ranging from 'no problems' to 'major problems'. The five dimensions can be summed into a health state, ranging from 0 to 100, with higher scores reflecting better health-related quality of life.
Healthcare utilisation by iMTA Medical Consumption Questionnaire (older adults) | baseline and after 6, 12 months
  The iMTA questionnaire is a questionnaire that measures healthcare utilisation and is often used in economic evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Gertrudis IJ Kempen, PhD, Study Chair — Maastricht University
Locations (1):
- MeanderGroep Zuid-Limburg, Landgraaf, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data and data dictionaries that underlie the results reported in articles that are published within this project are available from the corresponding author on reasonable request after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: Data will be available for researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to t.rooijackers@maastrichtuniversity.nl. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Metzelthin SF, Rooijackers TH, Zijlstra GAR, van Rossum E, Veenstra MY, Koster A, Evers SMAA, van Breukelen GJP, Kempen GIJM. Effects, costs and feasibility of the 'Stay Active at Home' Reablement training programme for home care professionals: study protocol of a cluster randomised controlled trial. BMC Geriatr. 2018 Nov 13;18(1):276. doi: 10.1186/s12877-018-0968-z. PMID 30424738
- [Background] Metzelthin SF, Zijlstra GA, van Rossum E, de Man-van Ginkel JM, Resnick B, Lewin G, Parsons M, Kempen GI. 'Doing with ...' rather than 'doing for ...' older adults: rationale and content of the 'Stay Active at Home' programme. Clin Rehabil. 2017 Nov;31(11):1419-1430. doi: 10.1177/0269215517698733. Epub 2017 Mar 14. PMID 29050508
- [Derived] Rooijackers TH, Metzelthin SF, van Rossum E, Kempen GIJM, Evers SMAA, Gabrio A, Zijlstra GAR. Economic Evaluation of a Reablement Training Program for Homecare Staff Targeting Sedentary Behavior in Community-Dwelling Older Adults Compared to Usual Care: A Cluster Randomized Controlled Trial. Clin Interv Aging. 2021 Dec 22;16:2095-2109. doi: 10.2147/CIA.S341221. eCollection 2021. PMID 35221681
- [Derived] Rooijackers TH, Zijlstra GAR, van Rossum E, Vogel RGM, Veenstra MY, Kempen GIJM, Metzelthin SF. Process evaluation of a reablement training program for homecare staff to encourage independence in community-dwelling older adults. BMC Geriatr. 2021 Jan 6;21(1):5. doi: 10.1186/s12877-020-01936-7. PMID 33407189